CLINICAL TRIAL: NCT05940428
Title: A Multicenter, Non-Randomized, Open-Label, Multiple-Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of ASKG712 Following Intravitreal Administration in Patients With Diabetic Macular Edema
Brief Title: A Study of ASKG712 in Patients With Diabetic Macular Edema
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Suzhou Aosaikang Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASKG712-CT-I-2
Record Dates: First submitted 2023-05-11; First posted 2023-07-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASKG712 (Experimental): Multiple doses of ASKG712 by intravitreal injection
  Interventions: Biological: ASKG712

INTERVENTIONS:
Biological: ASKG712 — ASKG712 is a recombinant anti-VEGF humanized monoclonal antibody and Ang-2 antagonist peptide fusion protein, which has high specificity for the binding of VEGF-A and Ang-2.
  Other Names: AM712

SUMMARY:
This multicenter, non-randomized, open-label, multiple-dose-escalation and dose-expansion study will investigate the safety, tolerability, pharmacokinetics and efficacy of ASKG712 following intravitreal administration in patients with diabetic macular edema (DME).

DETAILED DESCRIPTION:
The Part 1 of study is a multicenter, open-label, sequentially, multiple-dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and efficacy of ASKG712 in patients with DME. Patients will be sequentially enrolled into four different dose-level cohorts following accelerated titration combined with the traditional "3+3" design.

The Part 2 of study is a multicenter, open-label, sequentially, dose-expansion study to evaluate the safety, tolerability, pharmacokinetics and efficacy of ASKG712 in patients with DME.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of diabetes mellitus (Type 1 or Type 2)
2. Hemoglobin A1c of less than or equal to 12%
3. For women of childbearing potential: agreement to use acceptable contraceptive methods during the treatment period and for at least 90 days after the final dose of study treatment
4. Ability and willingness to undertake all scheduled visits and assessments
5. Macular thickening secondary to DME involving the center of the fovea
6. Decreased visual acuity attributable primarily to DME

Exclusion Criteria:

1. History of allergy or current allergic response to ASKG712 or fluorescein
2. Diseases that affect intravenous injection and venous blood sampling
3. Uncontrolled blood pressure
4. Systemic autoimmune diseases
5. Previous anti-VEGF drug treatment
6. Currently pregnant or breastfeeding, or intend to become pregnant during the study
7. Any uncontrolled clinical disorders
8. Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye
9. History of intraocular or periocular corticosteroid treatment in the study eye
10. Uncontrolled previous or current glaucoma in the study eye
11. Previous intraocular operations in the study eye
12. Active intraocular or periocular infection or active intraocular inflammation in the study eye
13. History of uveitis in either eye
14. Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of ocular adverse events (AEs) of the study eyes | 24 weeks
  Any relevant ocular observations derived from best corrected visual acuity (BCVA), intraocular pressure, slitlamp examination, ophthalmoscopy, optical coherence tomography (OCT), fundus photography, and angiography
2. Incidence of non-ocular AEs | 24 weeks
  Any clinical safety observations assessed by physical examination, vital signs, electrocardiograph (ECG) and clinical laboratory tests

SECONDARY OUTCOMES:
1. Area under the concentration time curve (AUC) | 24 weeks
  To evaluate the systemic pharmacokinetics of ASKG712 in patients with DME
2. Maximum plasma concentration (Cmax) | 24 weeks
  To evaluate the systemic pharmacokinetics of ASKG712 in patients with DME
3. Incidence of Anti-Drug Antibody (ADA) | 24 weeks
  To evaluate the immunogenicity of ASKG712 in patients with DME
4. Change From Baseline in BCVA in the Study Eye Over Time | 24 weeks
  To evaluate the efficacy of ASKG712 in patients with DME

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD or supporting information available